CLINICAL TRIAL: NCT05506137
Title: Xerostomia in Patients With a Life-limiting Condition or Frailty: a Double-blind Placebo-controlled Randomized Clinical Trial
Brief Title: Xerostomia in Patients With a Life-limiting Condition or Frailty
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-501084-41-00
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Xerostomia; Dry Mouth
Keywords: Xerostomia; Dry mouth; Pilocarpine
MeSH Terms: conditions — Xerostomia | interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: Pilocarpine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pilocarpine — study whether topical pilocarpine drops induce a clinically significant improvement in xerostomia
  Arms: Treatment
Other: Placebo — study whether topical pilocarpine drops induce a clinically significant improvement in xerostomia
  Arms: Placebo

SUMMARY:
Xerostomia, the subjective feeling of dry mouth, is a common symptom during the last year of life in patients with a life-limiting condition or frailty. Xerostomia leads to functional alterations (such as burning sensations, an altered taste perception, and difficulties with chewing, swallowing, and speaking), has disabling social consequences and significantly downgrades the perceived quality of life. It is an under-exposed and under-treated symptom often caused by alterations in the quality and quantity of saliva.

Locally administered pilocarpine could be a promising drug in this regard as it alleviates xerostomia by increasing the production of saliva.

ELIGIBILITY:
Inclusion Criteria:

* have a life-limiting condition or frailty
* have the complaint dry mouth ≥ 5 on an 11 point numerical rating scale (ranging from 0= no dry mouth to 10= worst dry mouth ever)
* fulfil the single SQ 'Would I be surprised if my patient dies within the year? (no)

Exclusion Criteria:

* their life expectancy is less than 4 weeks (the primary endpoint at 4 weeks)
* they have had radiotherapy to the salivary glands or suffer from Sjögrens disease (impact on dry mouth)
* cognitively impaired to such an extent that there is insufficient understanding to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The percentage responders at week 4 of topical pilocarpine administration, as compared to baseline. | 4 weeks
  A patient counts as a responder with, at least, a 2-point reduction on the 11-point NRS

SECONDARY OUTCOMES:
Mean difference in NRS dry mouth scores in the pilocarpine group at all time-points, as compared to the placebo group | 4 - 12 weeks
  Mean difference in NRS dry mouth scores is determined as mean change from baseline
Change in Oral Health-Related Quality of Life (OHRQoL) upon pilocarpine treatment, as compared to the placebo group | 4 - 12 weeks
  The OHRQoL is measured using the Geriatric Oral Health Assessment Index (GOHAI-NL)
Change in the Health-Related Quality of Life upon pilocarpine treatment, as compared to the placebo group | 4 - 12 weeks
  The HRQoL will be assessed using the EQ-5D-5L questionnaire
Change in clinical functioning upon pilocarpine treatment, as compared to the placebo group | 4 - 12 weeks
  Clinical functioning is determined using the Patient-reported functional status (PRFS) questionnaire
Change in the Global Perceived Effect (GPE) upon pilocarpine treatment, as compared to the placebo group | 4 - 12 weeks
  The GPE is determined by a globally experienced effect score
The durability of the effect of the use of pilocarpine on xerostomia | 4 - 12 weeks
  The durability will be displayed in percentage
The adherence rate of patients | 4 -12 weeks
  Adherence will be displayed in percentage
Possible side effects related to the intake of pilocarpine medication, as compared to the placebo group | 4 - 12 weeks
  Side effects are made transparent by providing an overview of which and how many side effects occur
Cost Effectiveness Analysis (CEA) of the pilocarpine treatment | 4 - 12 weeks
  The costst of patients is analysed using the medical consumption questionnaire (iMCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Marieke van den Beuken- van Everdingen, Prof., Principal Investigator — Maastricht University and/or Maastricht UMC+

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Theunissen M, Rideaux-Seferina S, Magdelijns FJ, Janssen DJA, van den Beuken-van Everdingen MHJ. Local Oral Pilocarpine Drops for Relieving Xerostomia (Dry Mouth) in the Elderly: A Pilot Study. J Am Med Dir Assoc. 2021 Jan;22(1):185-186. doi: 10.1016/j.jamda.2020.06.036. Epub 2020 Aug 13. No abstract available. PMID 32800514
- [Derived] van der Meulen AI, Neis EPJG, de Nijs EJM, Coenegracht BJEG, Stoppelenburg A, van den Beuken-van Everdingen MHJ, van der Linden YM. Dry mouth in patients with a life-limiting condition or frailty: a study protocol for two intervention studies and a nested qualitative sub-study (the Dry mOuth Project, DROP). BMC Palliat Care. 2023 Aug 23;22(1):120. doi: 10.1186/s12904-023-01242-0. PMID 37612654
- See also: ZonMW Programma Palliantie — https://www.zonmw.nl/nl/over-zonmw/onderwijs/programmas/project-detail/palliantie-meer-dan-zorg/dry-mouth-in-patients-with-a-life-limiting-condition-or-frailty-a-two-track-non-pharmacological-and/